CLINICAL TRIAL: NCT04439994
Title: Activation of Plasma miRNA and Proteins as a Result of Acute Experimental Pain
Brief Title: Activation of miRNA and Proteins After Acute Experimental Pain. (miRNA: Micro RNA)
Acronym: miRNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Assistant Professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20200015
Record Dates: First submitted 2020-06-16; First posted 2020-06-19 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Hypertonic Saline; Isotonic Saline
MeSH Terms: interventions — Saline Solution, Hypertonic; Sodium Chloride; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: two groups of subjects: one group will receive hypertonic injection (0.1 ml) and the other group will receive isotonic saline injection (0.1 ml)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertonic saline (Active Comparator): Each participant will be given i.d. in 0.1 mL volumes of a hypertonic saline solution. The subject will be blinded to the hypertonic/isotonic administration.
  Interventions: Other: hypertonic saline; Procedure: Blood sampling
- Isotonic Saline (Placebo Comparator): Each participant will be given i.d. in 0.1 mL volumes of a isotonic saline solution. The subject will be blinded to the hypertonic/isotonic administration.
  Interventions: Other: Saline injection; Procedure: Blood sampling

INTERVENTIONS:
Other: hypertonic saline — The participant will be given i.d. in 0.1 mL volumes of a hypertonic saline solution
  Arms: Hypertonic saline
Other: Saline injection — The participant will be given i.d. in 0.1 mL volumes of a saline solution
  Arms: Isotonic Saline
Procedure: Blood sampling — Whole blood samples (5 mL per each time point, a total of 20 mL per subject) will be collected

SUMMARY:
In this experiment, the investigators would like to test the following:

1. Does acute pain induced by hypertonic injection cause changes in plasma miRNA and protein expression ?
2. Can these canges correlate with the development of local hyperalgesia?
3. How does the plasma miRNA expression change over a duration of 24 hours post pain induction ?
4. Which mRNA targets are potentially affected by acute pain?

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women in the age 18-80 years
* Speak and understand English

Exclusion Criteria:

* Acute and chronic pain
* Pregnancy or breastfeeding
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Present or previous history of neurological, dermatological, immunological, musculoskeletal, cardiac disorder or mental illnesses that may affect the results (e.g. Neuropathy, muscular pain in the upper extremities, etc.)
* Lack of ability to cooperate
* Current use of medications that may affect the trial, such as antipsychotics and pain killers as well as systemic or topical steroids and anti-inflammatory drugs.
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
miRNA expression over time | Before injection
  Plasma miRNA evaluation
miRNA expression over time | 30 minutes post-injection
  Plasma miRNA evaluation
miRNA expression over time | 3 hours post-injection
  Plasma miRNA evaluation
miRNA expression over time | 24 hours post-injection
  Plasma miRNA evaluation
Protein expression over time | Before injection
  Plasma protein evaluation
Protein expression over time | 30 minutes post-injection
  Plasma protein evaluation
Protein expression over time | 3 hours post-injection
  Plasma protein evaluation
Protein expression over time | 24 hours post-injection
  Plasma protein evaluation

SECONDARY OUTCOMES:
Assessment of pain: visual analog scale | 20 minutes
  Pain following capsaicin injection will be monitored for 20 minutes using a computerized 100 mm visual analog scale (eVAS software Aalborg University, Denmark), installed on a tablet.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aalborg University, Aalborg, North Denmark
  - AAlborg University, Aalborg, North Denmark

REFERENCES:
- [Derived] Giordano R, Gerra MC, Okutani H, Lo Vecchio S, Stensballe A, Petersen KK, Arendt-Nielsen L. The temporal expression of circulating microRNAs after acute experimental pain in humans. Eur J Pain. 2023 Mar;27(3):366-377. doi: 10.1002/ejp.2062. Epub 2022 Dec 9. PMID 36453122